CLINICAL TRIAL: NCT07232576
Title: A Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of SHR-1139 in Patients With moderate-to- Severe Active Ulcerative Colitis.
Brief Title: A Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of SHR-1139 in Patients With Moderate-to-severe Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1139-202
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Adult Patients With Moderately to Severely Active Ulcerative Colitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental): SHR-1139 Injection
  Interventions: Drug: SHR-1139 intravenous injection.

INTERVENTIONS:
Drug: SHR-1139 intravenous injection. — SHR-1139 intravenous injection.

SUMMARY:
This phase 2 study is being conducted to evaluate the efficacy, safety and pharmacokinetics of SHR-1139 in patients with moderate to severe active ulcerative colitis.

This study consists 2 treatment parts, the Induction treatment part and Maintenance treatment part. The periods of Induction treatment part and Maintenance treatment part are 12 weeks and 48 weeks separately.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subject age ≥ 18 and ≤ 75 years of age at screening.
2. the body mass index (BMI= weight (kg)/height (2 m ²)) of the subjects is ≥ 18 kg/m ² at the screening.
3. Subject has active Ulcerative Colitis with a 9-point modified Mayo score of 4-9 at baseline, with an endoscopic subscore of ≥ 2 (confirmed by central read). (NOTE: endoscopy should be performed within 14 days prior to baseline visit), and rectal bleeding subscore of ≥1.
4. Subject has at least a 90-days history of Ulcerative Colitis diagnosis at baseline.
5. Subject is deemed by the physician as having inadequate response, loss of response or intolerance (Appendix 5) to at least one conventional treatment (oral 5-ASA, immunosuppressants or corticosteroids), or was previously exposed to anti-TNF therapy (e.g., infliximab, adalimumab) or other biological treatment.
6. Subject is capable of providing a signed and dated informed consent form indicating the subject has been informed of all pertinent aspects of the study.
7. All women of childbearing potential and their male partners must commit to using at least two methods of contraception with one method being highly effective throughout the duration of the study, and for 72 weeks after last dose of study medication.

Exclusion Criteria:

1. Subject has a diagnosis of indeterminate colitis, or clinical findings suggestive of Crohn's Disease.
2. Subject with Ulcerative Colitis, which is confined to a proctitis (distal 15 cm or less).
3. Treatment naïve subject diagnosed with Ulcerative Colitis (without previous exposure to any of the following therapies for UC treatment: oral 5-ASA, corticosteroids, immunosuppressants, or biological treatments).
4. Subject is displaying clinical signs of ischemic colitis, fulminant colitis or toxic megacolon.
5. Subject had previous surgery as a treatment for Ulcerative Colitis or likely to require surgery during the study period.
6. Screening endoscopic examination revealed that the subjects had a history of gastrointestinal dysplasia (atypical hyperplasia)/cancer or dysplasia (atypical hyperplasia)/cancer. Except for completely resected low-grade dysplasia.
7. Subject has evidence of pathogenic bowel infection. Subjects had Clostridium difficile or other intestinal infection within 30 days of screening endoscopy or test positive at screening for C. difficile toxin or other intestinal pathogens.
8. Subject currently has or had:

   8.1 A clinically significant infection within 1 month of baseline (e.g., those requiring hospitalization or parenteral antimicrobial therapy or have opportunistic infections).

   8.2 A history of more than one episode of herpes zoster, or disseminated zoster (single episode).

   8.3 Any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the study.

   8.4 Any infection requiring antimicrobial therapy within 2 weeks of screening.
9. Subject is receiving any of the following therapies:

9.1 Cyclosporine, mycophenolate, tacrolimus、JAK inhibitors within 4 weeks prior to baseline.

9.2 Interferon therapy within 8 weeks prior to baseline. 9.3 Intravenous corticosteroids or rectally administered formulation of corticosteroids or 5-ASA within 2 weeks prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve clinical response (based on modified Mayo score) at week 12. | at week 12.

SECONDARY OUTCOMES:
The proportion of subjects who achieve clinical remission (based on modified Mayo score) at week 12 and week 60. | at week 12 and week 60.
The proportion of subjects who achieve endoscopic improvement, endoscopic remission and systemic remission at week 12 and week 60. | at week 12 and week 60.
The proportion of subjects who achieve clinical response (based on modified Mayo score) at week 60. | at week 12 and week 60.
The proportion of subjects whose partial Mayo score ≤1 at each visit. | at week 4, 8, 12, 22, 36, 42 and week 60.
The proportion of subjects whose total Mayo score ≤2 and no individual sub-score >1 at week 12 and week 60. | at week 12 and week 60.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital,Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided